CLINICAL TRIAL: NCT02499471
Title: Brown Adipose Tissue Activity and Thyroid Hormone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL 39146.068.11
Record Dates: First submitted 2015-07-06; First posted 2015-07-16 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Hypothyroidism; Hyperthyroidism; Obesity
MeSH Terms: conditions — Hypothyroidism; Hyperthyroidism; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Before levothyroxine therapy 137.75 μg (Other): 18F-FDG PET CT scan after mild cold exposure 6.8 ± 2.8 weeks after thyroidectomy, when plasma free T4-levels were at the minimum, before daily levothyroxine therapy 137.75 ± 25.75 μg.
  Interventions: Other: Levothyroxine therapy (137.75 ± 23.75 μg/day)
- After levothyroxine therapy 137.75 μg (Other): 18F-FDG PET CT scan after mild cold exposure four to six months after the initial measurements, after daily levothyroxine therapy 137.75 μg (fT4 levels 23.1 ± 3.9 pmol/L, TSH 0.5 ± 0.6 mU/L)
  Interventions: Other: Levothyroxine therapy (137.75 ± 23.75 μg/day)

INTERVENTIONS:
Other: Levothyroxine therapy (137.75 ± 23.75 μg/day) — This study was a longitudinal study in an academic center, with a follow-up period of 6 months. Ten patients with well-differentiated thyroid carcinoma eligible for surgical treatment and subsequent radioactive iodine ablation therapy were studied in a hypothyroid state after thyroidectomy and in a subclinical hyperthyroid state (TSH-suppression according to standard treatment protocol).

SUMMARY:
Rationale: During the last decades, research in possible therapies for existing obesity and developmental factors causing obesity has explosively increased. Recently renewed interest aroused for a tissue playing a possible role in both development and therapy for obesity: brown adipose tissue (BAT).

To define the relation between BAT and thyroid hormone, the investigators set up the following research protocol. In this protocol BAT activity will be determined in subjects that underwent thyroidectomy for well-differentiated thyroid carcinoma.

Objective: To study the effect of thyroid hormone and thyroid-stimulating hormone on brown adipose tissue activity.

Study design: Determine BAT activity after thyroidectomy in well-differentiated thyroid carcinoma patients.

Study population: Patients that underwent thyroidectomy for well-differentiated thyroid carcinoma, male and female, aged 18-65 years.

Intervention: FDG-PET-CT-imaging ([18F]fluorodeoxyglucose positron-emission-tomography computed-tomography) of BAT activity will be performed under cold stimulation twice.

For patients clinically withdrawn from thyroid hormone suppletion, the first occasion will be in a hypothyroid state within 4-6 weeks after thyroidectomy and the second measurement will take place in a euthyroid state 4 months after the start of thyroid hormone treatment.

For patients receiving recombinant-thyroid-stimulating-hormone injections, the first occasion will be shortly after the injection in a state of high thyroid-stimulating hormone levels. The second measurement will be in a euthyroid state 4 months after the injection.

Main study parameters/endpoints: The main endpoint of this study is the effect of thyroid hormone and thyroid-stimulating hormone on BAT activity in kBq (kilobecquerel) and SUV (standard uptake value). Secondary endpoints are the effects of thyroid hormone and thyroid-stimulating hormone on energy metabolism, body core temperature, skin surface temperatures and skin perfusion.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The absorbed radiation dose from the FDG PET-CT scan after administration of 74 MBq (megabecquerel) of 18F-FDG is 2.8 mSv (miliSievert).

ELIGIBILITY:
Inclusion Criteria:

* Male or postmenopausal females undergoing a total thyroidectomy for well-differentiated thyroid carcinoma
* Age 18-65 years
* Stable physical activity levels for at least six months
* Note: In case of use of anticoagulation, the dose will be adjusted according to plasma thyroid hormone values.

Exclusion Criteria:

* Psychologically unstable subjects (as judged by the treating medical specialist)
* Subjects with mental retardation (as judged by the treating medical specialist)
* Subjects with severe behavior disorders (as judged by the treating medical specialist)
* Pregnant subjects
* The use of the following medication is an exclusion criterium; ß-blockers
* Participation in an intensive weight-loss program or vigorous exercise program during the last year before the start of the study
* Abuse of drugs and/or alcohol
* Severe diabetes which requires application of insulin or patients with diabetes-related complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Cold-induced brown adipose tissue activity | 1 day
  Measured with 18FDG PET/CT scan after personalised cooling protocol

SECONDARY OUTCOMES:
Energy expenditure | 1 day
  Energy expenditure measured with ventilated hood system
Body core temperature | 1 day
  Body core temperature measured with CorTemp telemetric pill
Skin temperatures | 1 day
  Skin temperatures measured with iButton wireless dataloggers at 14 ISO-defined positions on the skin
Skin perfusion | 1 day
  Skin perfusion measured with laser-doppler flowmetry on hand and forearm

CONTACTS AND LOCATIONS:
Overall Officials: Wouter van Marken Lichtenbelt, Professor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Mokdad AH, Marks JS, Stroup DF, Gerberding JL. Actual causes of death in the United States, 2000. JAMA. 2004 Mar 10;291(10):1238-45. doi: 10.1001/jama.291.10.1238. PMID 15010446
- [Background] van Marken Lichtenbelt WD, Vanhommerig JW, Smulders NM, Drossaerts JM, Kemerink GJ, Bouvy ND, Schrauwen P, Teule GJ. Cold-activated brown adipose tissue in healthy men. N Engl J Med. 2009 Apr 9;360(15):1500-8. doi: 10.1056/NEJMoa0808718. PMID 19357405
- [Background] Virtanen KA, Lidell ME, Orava J, Heglind M, Westergren R, Niemi T, Taittonen M, Laine J, Savisto NJ, Enerback S, Nuutila P. Functional brown adipose tissue in healthy adults. N Engl J Med. 2009 Apr 9;360(15):1518-25. doi: 10.1056/NEJMoa0808949. PMID 19357407
- [Background] Cannon B, Nedergaard J. Brown adipose tissue: function and physiological significance. Physiol Rev. 2004 Jan;84(1):277-359. doi: 10.1152/physrev.00015.2003. PMID 14715917
- [Background] Saito M, Okamatsu-Ogura Y, Matsushita M, Watanabe K, Yoneshiro T, Nio-Kobayashi J, Iwanaga T, Miyagawa M, Kameya T, Nakada K, Kawai Y, Tsujisaki M. High incidence of metabolically active brown adipose tissue in healthy adult humans: effects of cold exposure and adiposity. Diabetes. 2009 Jul;58(7):1526-31. doi: 10.2337/db09-0530. Epub 2009 Apr 28. PMID 19401428
- [Background] Orava J, Nuutila P, Lidell ME, Oikonen V, Noponen T, Viljanen T, Scheinin M, Taittonen M, Niemi T, Enerback S, Virtanen KA. Different metabolic responses of human brown adipose tissue to activation by cold and insulin. Cell Metab. 2011 Aug 3;14(2):272-9. doi: 10.1016/j.cmet.2011.06.012. PMID 21803297
- [Background] van der Lans AA, Hoeks J, Brans B, Vijgen GH, Visser MG, Vosselman MJ, Hansen J, Jorgensen JA, Wu J, Mottaghy FM, Schrauwen P, van Marken Lichtenbelt WD. Cold acclimation recruits human brown fat and increases nonshivering thermogenesis. J Clin Invest. 2013 Aug;123(8):3395-403. doi: 10.1172/JCI68993. Epub 2013 Jul 15. PMID 23867626
- [Background] TATA JR, ERNSTER L, LINDBERG O. Control of basal metabolic rate by thyroid hormones and cellular function. Nature. 1962 Mar 17;193:1058-60. doi: 10.1038/1931058a0. No abstract available. PMID 13919771
- [Background] Goglia F, Silvestri E, Lanni A. Thyroid hormones and mitochondria. Biosci Rep. 2002 Feb;22(1):17-32. doi: 10.1023/a:1016056905347. PMID 12418548
- [Background] Bianco AC, Salvatore D, Gereben B, Berry MJ, Larsen PR. Biochemistry, cellular and molecular biology, and physiological roles of the iodothyronine selenodeiodinases. Endocr Rev. 2002 Feb;23(1):38-89. doi: 10.1210/edrv.23.1.0455. PMID 11844744
- [Background] Johannsen DL, Galgani JE, Johannsen NM, Zhang Z, Covington JD, Ravussin E. Effect of short-term thyroxine administration on energy metabolism and mitochondrial efficiency in humans. PLoS One. 2012;7(7):e40837. doi: 10.1371/journal.pone.0040837. Epub 2012 Jul 26. PMID 22844412
- [Background] Lee JY, Takahashi N, Yasubuchi M, Kim YI, Hashizaki H, Kim MJ, Sakamoto T, Goto T, Kawada T. Triiodothyronine induces UCP-1 expression and mitochondrial biogenesis in human adipocytes. Am J Physiol Cell Physiol. 2012 Jan 15;302(2):C463-72. doi: 10.1152/ajpcell.00010.2011. Epub 2011 Nov 9. PMID 22075692
- [Background] de Jesus LA, Carvalho SD, Ribeiro MO, Schneider M, Kim SW, Harney JW, Larsen PR, Bianco AC. The type 2 iodothyronine deiodinase is essential for adaptive thermogenesis in brown adipose tissue. J Clin Invest. 2001 Nov;108(9):1379-85. doi: 10.1172/JCI13803. PMID 11696583
- [Background] Endo T, Kobayashi T. Thyroid-stimulating hormone receptor in brown adipose tissue is involved in the regulation of thermogenesis. Am J Physiol Endocrinol Metab. 2008 Aug;295(2):E514-8. doi: 10.1152/ajpendo.90433.2008. Epub 2008 Jun 17. PMID 18559984
- [Background] Lopez M, Varela L, Vazquez MJ, Rodriguez-Cuenca S, Gonzalez CR, Velagapudi VR, Morgan DA, Schoenmakers E, Agassandian K, Lage R, Martinez de Morentin PB, Tovar S, Nogueiras R, Carling D, Lelliott C, Gallego R, Oresic M, Chatterjee K, Saha AK, Rahmouni K, Dieguez C, Vidal-Puig A. Hypothalamic AMPK and fatty acid metabolism mediate thyroid regulation of energy balance. Nat Med. 2010 Sep;16(9):1001-8. doi: 10.1038/nm.2207. Epub 2010 Aug 29. PMID 20802499
- [Background] Andersen S, Kleinschmidt K, Hvingel B, Laurberg P. Thyroid hyperactivity with high thyroglobulin in serum despite sufficient iodine intake in chronic cold adaptation in an Arctic Inuit hunter population. Eur J Endocrinol. 2012 Mar;166(3):433-40. doi: 10.1530/EJE-11-0888. Epub 2011 Dec 14. PMID 22170797
- [Background] Louzada RA, Santos MC, Cavalcanti-de-Albuquerque JP, Rangel IF, Ferreira AC, Galina A, Werneck-de-Castro JP, Carvalho DP. Type 2 iodothyronine deiodinase is upregulated in rat slow- and fast-twitch skeletal muscle during cold exposure. Am J Physiol Endocrinol Metab. 2014 Dec 1;307(11):E1020-9. doi: 10.1152/ajpendo.00637.2013. Epub 2014 Oct 7. PMID 25294216
- [Background] Lahesmaa M, Orava J, Schalin-Jantti C, Soinio M, Hannukainen JC, Noponen T, Kirjavainen A, Iida H, Kudomi N, Enerback S, Virtanen KA, Nuutila P. Hyperthyroidism increases brown fat metabolism in humans. J Clin Endocrinol Metab. 2014 Jan;99(1):E28-35. doi: 10.1210/jc.2013-2312. Epub 2013 Dec 20. PMID 24152690
- [Background] van Marken Lichtenbelt WD, Daanen HA, Wouters L, Fronczek R, Raymann RJ, Severens NM, Van Someren EJ. Evaluation of wireless determination of skin temperature using iButtons. Physiol Behav. 2006 Jul 30;88(4-5):489-97. doi: 10.1016/j.physbeh.2006.04.026. Epub 2006 Jun 23. PMID 16797616
- [Background] Kingma BR, Frijns AJ, Saris WH, van Steenhoven AA, Lichtenbelt WD. Increased systolic blood pressure after mild cold and rewarming: relation to cold-induced thermogenesis and age. Acta Physiol (Oxf). 2011 Dec;203(4):419-27. doi: 10.1111/j.1748-1716.2011.02336.x. Epub 2011 Aug 12. PMID 21707931
- [Background] Vosselman MJ, van der Lans AA, Brans B, Wierts R, van Baak MA, Schrauwen P, van Marken Lichtenbelt WD. Systemic beta-adrenergic stimulation of thermogenesis is not accompanied by brown adipose tissue activity in humans. Diabetes. 2012 Dec;61(12):3106-13. doi: 10.2337/db12-0288. Epub 2012 Aug 7. PMID 22872233
- [Result] Skarulis MC, Celi FS, Mueller E, Zemskova M, Malek R, Hugendubler L, Cochran C, Solomon J, Chen C, Gorden P. Thyroid hormone induced brown adipose tissue and amelioration of diabetes in a patient with extreme insulin resistance. J Clin Endocrinol Metab. 2010 Jan;95(1):256-62. doi: 10.1210/jc.2009-0543. Epub 2009 Nov 6. PMID 19897683
- [Result] Danforth E Jr, Burger A. The role of thyroid hormones in the control of energy expenditure. Clin Endocrinol Metab. 1984 Nov;13(3):581-95. doi: 10.1016/s0300-595x(84)80039-0. PMID 6391756
- [Result] BARKER SB, KLITGAARD HM. Metabolism of tissues excised from thyroxine-injected rats. Am J Physiol. 1952 Jul;170(1):81-6. doi: 10.1152/ajplegacy.1952.170.1.81. No abstract available. PMID 12985867
- [Result] Nedergaard J, Golozoubova V, Matthias A, Asadi A, Jacobsson A, Cannon B. UCP1: the only protein able to mediate adaptive non-shivering thermogenesis and metabolic inefficiency. Biochim Biophys Acta. 2001 Mar 1;1504(1):82-106. doi: 10.1016/s0005-2728(00)00247-4. PMID 11239487
- [Result] Kim MS, Hu HH, Aggabao PC, Geffner ME, Gilsanz V. Presence of brown adipose tissue in an adolescent with severe primary hypothyroidism. J Clin Endocrinol Metab. 2014 Sep;99(9):E1686-90. doi: 10.1210/jc.2014-1343. Epub 2014 Jun 10. PMID 24915119
- [Result] Bilezikian JP, Loeb JN. The influence of hyperthyroidism and hypothyroidism on alpha- and beta-adrenergic receptor systems and adrenergic responsiveness. Endocr Rev. 1983 Fall;4(4):378-88. doi: 10.1210/edrv-4-4-378. PMID 6317368
- [Result] Castillo M, Hall JA, Correa-Medina M, Ueta C, Kang HW, Cohen DE, Bianco AC. Disruption of thyroid hormone activation in type 2 deiodinase knockout mice causes obesity with glucose intolerance and liver steatosis only at thermoneutrality. Diabetes. 2011 Apr;60(4):1082-9. doi: 10.2337/db10-0758. Epub 2011 Feb 18. PMID 21335378
- [Result] Silva JE, Bianco SD. Thyroid-adrenergic interactions: physiological and clinical implications. Thyroid. 2008 Feb;18(2):157-65. doi: 10.1089/thy.2007.0252. PMID 18279016
- [Result] Volzke H, Alte D, Dorr M, Wallaschofski H, John U, Felix SB, Rettig R. The association between subclinical hyperthyroidism and blood pressure in a population-based study. J Hypertens. 2006 Oct;24(10):1947-53. doi: 10.1097/01.hjh.0000244942.57417.8e. PMID 16957553
- [Result] Liu D, Jiang F, Shan Z, Wang B, Wang J, Lai Y, Chen Y, Li M, Liu H, Li C, Xue H, Li N, Yu J, Shi L, Bai X, Hou X, Zhu L, Lu L, Wang S, Xing Q, Teng W. A cross-sectional survey of relationship between serum TSH level and blood pressure. J Hum Hypertens. 2010 Feb;24(2):134-8. doi: 10.1038/jhh.2009.44. Epub 2009 Jun 25. PMID 19554027
- [Result] Thrush AB, Gagnon A, Sorisky A. PKC activation is required for TSH-mediated lipolysis via perilipin activation. Horm Metab Res. 2012 Oct;44(11):825-31. doi: 10.1055/s-0032-1316332. Epub 2012 Jun 22. PMID 22730012
- [Result] Gagnon A, Antunes TT, Ly T, Pongsuwan P, Gavin C, Lochnan HA, Sorisky A. Thyroid-stimulating hormone stimulates lipolysis in adipocytes in culture and raises serum free fatty acid levels in vivo. Metabolism. 2010 Apr;59(4):547-53. doi: 10.1016/j.metabol.2009.08.018. Epub 2009 Oct 20. PMID 19846175
- [Result] Bartelt A, Bruns OT, Reimer R, Hohenberg H, Ittrich H, Peldschus K, Kaul MG, Tromsdorf UI, Weller H, Waurisch C, Eychmuller A, Gordts PL, Rinninger F, Bruegelmann K, Freund B, Nielsen P, Merkel M, Heeren J. Brown adipose tissue activity controls triglyceride clearance. Nat Med. 2011 Feb;17(2):200-5. doi: 10.1038/nm.2297. Epub 2011 Jan 23. PMID 21258337
- [Result] Cannon B, Nedergaard J. Thyroid hormones: igniting brown fat via the brain. Nat Med. 2010 Sep;16(9):965-7. doi: 10.1038/nm0910-965. No abstract available. PMID 20823876
- [Derived] Broeders EP, Vijgen GH, Havekes B, Bouvy ND, Mottaghy FM, Kars M, Schaper NC, Schrauwen P, Brans B, van Marken Lichtenbelt WD. Thyroid Hormone Activates Brown Adipose Tissue and Increases Non-Shivering Thermogenesis--A Cohort Study in a Group of Thyroid Carcinoma Patients. PLoS One. 2016 Jan 19;11(1):e0145049. doi: 10.1371/journal.pone.0145049. eCollection 2016. PMID 26784028